CLINICAL TRIAL: NCT02705001
Title: Nurse Graduateness and Patient Outcomes: a Cross Sectional Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Weill Cornell Medical College in Qatar (Other); University of Hull (Other); Australian Catholic University (Other); University of South Australia (Other)
Responsible Party: Principal Investigator, Dr. Richard Gray, Executive Director of Nursing, Research, Hamad Medical Corporation
Other Study IDs: 15363/15
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: no Spedific Condition, All-cause In-patient Mortality
MeSH Terms: interventions — Emergency Service, Hospital

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: all admissions except accident and emergency — No additional intervention, retrospective study

SUMMARY:
This research project is relevant to the identification of the relationship, and its significance, between patient morality and a number of demographic, clinical and corporate characteristics. Two separate data sets have been compiled linking the existing intervention and employment data, one focusing on the admitting nurse and another one considering all the nurses involved in each intervention. Several statistical experiments will take place to support or reject the main hypothesis: higher nurse education, satisfaction and staffing levels result to lower patient mortality.

DETAILED DESCRIPTION:
The primary research objective is to investigate the relationship between the education, satisfaction and staffing level of the nurses and the mortality rate across HMC. The relationship between mortality will be investigated against some additional demographic characteristics of the patient and the nurses as well as a umber of clinical parameters like the length of stay and the severity of the interventions. To achieve that data will be retrospectively collected from the Human Resources database containing the nurse education and demographic information and will combine it to the intervention data coming from the clinical information systems of all major public hospitals in Qatar excluding accident and emergency cases to avoid confounding. Rigorous statistical analysis will be conducted to obtain the significance of this relationship within expected confidence intervals. The end result of that process is to find whether there is a significant positive or negative relationship between nurse education and mortality rate.

For confounding purposes Accident and Emergency data have been excluded, we have performed several adjusted and unadjusted Logistic Regression tests and taking into consideration the clustering effect of the data.

ELIGIBILITY:
Exclusion Criteria:

* Accident and emergency patients
* Records with negative length of stay
* Records with incorrect patient demographics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients that visited the 7 participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1252 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
All-cause In-Patient Mortality | 6 months

IPD SHARING:
Plan to Share IPD: No